CLINICAL TRIAL: NCT03461289
Title: Phase 3, Open-Label, Single-Arm, Single-Dose Gene Replacement Therapy Clinical Trial for Patients With Spinal Muscular Atrophy Type 1 With One or Two SMN2 Copies Delivering AVXS-101 by Intravenous Infusion
Brief Title: Single-Dose Gene Replacement Therapy Clinical Trial for Participants With Spinal Muscular Atrophy Type 1
Acronym: STRIVE-EU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVXS-101-CL-302; 2017-000266-29 (EudraCT Number); COAV101A12301 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2018-03-04; First posted 2018-03-12 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: SMA
MeSH Terms: interventions — Zolgensma

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, single-dose, trial of onasemnogene abeparvovec-xioi
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Onasemnogene Abeparvovec-xioi (Experimental): Onasemnogene abeparvovec-xioi is a non-replicating recombinant adeno-associated virus serotype 9 (AAV9) containing the human survival motor neuron (SMN) gene under the control of the cytomegalovirus (CMV) enhancer/chicken β-actin-hybrid promoter (CB).
  Interventions: Biological: Onasemnogene Abeparvovec-xioi

INTERVENTIONS:
Biological: Onasemnogene Abeparvovec-xioi — Onasemnogene abeparvovec-xioi is a non-replicating recombinant adeno-associated virus serotype 9 (AAV9) containing the human survival motor neuron (SMN) gene under the control of the cytomegalovirus (CMV) enhancer/chicken β-actin-hybrid promoter (CB).
  Other Names: AVXS-101; OAV101; Zolgensma

SUMMARY:
Phase 3, open-label, single-arm, single-dose, trial of onasemnogene abeparvovec-xioi (gene replacement therapy) in patients with spinal muscular atrophy (SMA) Type 1 who meet enrollment criteria and are genetically defined by a biallelic pathogenic mutation of the survival motor neuron 1 gene (SMN1) with one or two copies of survival motor neuron 2 gene (SMN2). Up to 30 patients < 6 months (< 180 days) of age at the time of gene replacement therapy (Day 1) will be enrolled.

DETAILED DESCRIPTION:
Phase 3, open-label, single-arm, single-dose, trial of onasemnogene abeparvovec-xioi (gene replacement therapy) in patients with spinal muscular atrophy (SMA) Type 1 who meet enrollment criteria and are genetically defined by a biallelic pathogenic mutation of the survival motor neuron 1 gene (SMN1) with one or two copies of survival motor neuron 2 gene (SMN2). 30 patients < 6 months (< 180 days) of age at the time of gene replacement therapy (Day 1) will be enrolled.

The trial includes a screening period, a gene replacement therapy period, and a follow-up period. During the screening period (Days -30 to -2), patients whose parent(s)/legal guardian(s) provide informed consent will complete screening procedures to determine eligibility for trial enrollment. Patients who meet the entry criteria will enter the in-patient gene replacement therapy period (Day -1 to Day 3). On Day -1, patients will be admitted to the hospital for pre-treatment baseline procedures. On Day 1, patients will receive a one-time intravenous (IV) infusion of onasemnogene abeparvovec-xioi, and will undergo in-patient safety monitoring over the next 48 hours. Patients may be discharged 48 hours after the infusion, based on Investigator judgment. During the outpatient follow-up period (Days 4 to End of Trial at 18 months of age), patients will return at regularly scheduled intervals for efficacy and safety assessments until the End of Trial when the patient reaches 18 months of age. After the End of Trial visit, eligible patients will be asked to participate into the long-term follow up trial.

All post-treatment visits will be relative to the date on which gene replacement therapy is administered, until the patient is 14 months of age, after which they will be relevant to the patient's date of birth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SMA Type 1 as determined by diagnosis of SMA based on gene mutation analysis with biallelic SMN1 mutations (deletion or point mutations) and one or two copies of SMN2 [inclusive of the known SMN2 gene modifier mutation (c.859G>C)]
* Patients must be < 6 months (< 180 days) of age at the time of onasemnogene abeparvovec-xioi infusion
* Patients must have a swallowing evaluation test performed prior to administration of gene replacement therapy

Exclusion Criteria:

* Previous, planned or expected scoliosis repair surgery/procedure prior to 18 months of age
* Use of invasive ventilatory support (tracheotomy with positive pressure) or pulse oximetry < 95% saturation at screening
* Use or requirement of non-invasive ventilatory support for 12 or more hours daily in the two weeks prior to dosing
* Patient with signs of aspiration based on a swallowing test or whose weight-for-age falls below the 3rd percentile based on World Health Organization (WHO) Child Growth Standards and unwilling to use an alternative method to oral feeding
* Participation in recent SMA treatment clinical trial (with the exception of observational cohort studies or non-interventional studies) or receipt of an investigational or commercial compound, product or therapy administered with the intent to treat SMA (eg, nusinersen, valproic acid,) at any time prior to screening for this trial.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AveXis Medinfo, Study Chair — Sponsor GmbH
Locations (10):
- Belgium (2):
  - University Hospital Ghent Neuromuscular reference center, Ghent
  - Neuropédiatrie - Centre de Référence des Maladies Neuromusculaires, Liège
- Hôpital Armand Trousseau, Paris, France
- Italy (5):
  - Istituto Gianninia Gaslini, Genova
  - Policlinico "G. Martino", Messina
  - Carlo Besta Neurological Research Institute, Milan
  - University of Milan, Milan
  - Policlinico Gemelli, Rome
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - The John Walton Muscular Dystrophy Research Centre MRC Centre for Neuromuscular Diseases at Newcastle, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/.

REFERENCES:
- [Derived] Mercuri E, Muntoni F, Baranello G, Masson R, Boespflug-Tanguy O, Bruno C, Corti S, Daron A, Deconinck N, Servais L, Straub V, Ouyang H, Chand D, Tauscher-Wisniewski S, Mendonca N, Lavrov A; STR1VE-EU study group. Onasemnogene abeparvovec gene therapy for symptomatic infantile-onset spinal muscular atrophy type 1 (STR1VE-EU): an open-label, single-arm, multicentre, phase 3 trial. Lancet Neurol. 2021 Oct;20(10):832-841. doi: 10.1016/S1474-4422(21)00251-9. PMID 34536405
- [Derived] Day JW, Mendell JR, Mercuri E, Finkel RS, Strauss KA, Kleyn A, Tauscher-Wisniewski S, Tukov FF, Reyna SP, Chand DH. Clinical Trial and Postmarketing Safety of Onasemnogene Abeparvovec Therapy. Drug Saf. 2021 Oct;44(10):1109-1119. doi: 10.1007/s40264-021-01107-6. Epub 2021 Aug 12. PMID 34383289
- See also: The Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17805
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1068
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=528

RESULTS

PARTICIPANT FLOW:
Groups:
- Onasemnogene Abeparvovec-xioi: Participants received a single dose of onasemnogene abeparvovec-xioi administered as an intravenous (IV) infusion over 60 minutes at a dose of 1.1 × 10^14 vg/kg (vector genome per kilogram) on Day 1 of the overall study.
Period: Overall Study
Arm/Group | Onasemnogene Abeparvovec-xioi
Started | 33
Completed | 32
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Onasemnogene Abeparvovec-xioi
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.055 (1.2799)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 4
  Italy | 23
  United Kingdom | 4
  France | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieve Independent Sitting for at Least 10 Seconds
Description: Independent sitting is defined by the World Health Organization Multicentre Growth Reference Study, confirmed by video recording, as a participant who sits up straight with head erect for at least 10 seconds; participant does not use arms or hands to balance body or support position.
Time Frame: From Day 1 up to 18 Months of Age Visit (Up to a Maximum of Approximately 17 Months)
Population: The analysis population was the Intent-to-Treat (ITT) population which consisted of symptomatic participants with bi-allelic deletion of SMN1 (exon 7/8 common homozygous deletions) and 2 copies of SMN2 without the known gene modifier mutation (c.859G>C) who received an IV infusion of onasemnogene abeparvovec-xioi at less than 180 days of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Onasemnogene Abeparvovec-xioi
Number analyzed (Participants) | 32
Participants | 14

2. Secondary Outcome: Event-free Survival at 14 Months of Age
Description: Event-free survival at 14 months of age was defined as the number of participants who did not die, did not require permanent ventilation and did not withdraw from the study by 14 months of age.
Time Frame: Up to 14 months of age
Population: The analysis population was the ITT population which consisted of symptomatic participants with bi-allelic deletion of SMN1 (exon 7/8 common homozygous deletions) and 2 copies of SMN2 without the known gene modifier mutation (c.859G>C) who received an IV infusion of onasemnogene abeparvovec-xioi at less than 180 days of age.
Measure: Count of Participants; unit: Participants
Arm/Group | Onasemnogene Abeparvovec-xioi
Number analyzed (Participants) | 32
Participants | 31
Statistical Analysis 1: Comparison: Onasemnogene Abeparvovec-xioi; Test type: Superiority; p < 0.0001, Fisher Exact; Difference of Proportion = 0.71, 95% CI 2-sided [0.48 to 0.87]; Data for the current study were compared to historical control data (Finkel et al 2014 - PubMed 25080519) where 6 out of 23 (26.1%) babies were alive and did not need mechanical ventilation at 14 months of age

ADVERSE EVENTS:
Time Frame: From Day 1 up to 30 days after the 18 months of age visit (up to a maximum of 17 months)
Description: Non-serious treatment emergent AEs were collected from Day 1 until 18 months of age visit.
Arm/Group | Onasemnogene Abeparvovec-xioi
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 19/33
Other Adverse Events (participants affected / at risk) | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onasemnogene Abeparvovec-xioi (N=33)
Gastrostomy (Surgical and medical procedures) | 2 (3)
Hospitalisation (Surgical and medical procedures) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Coagulation test abnormal (Investigations) | 1 (1)
Pulmonary function test (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (2)
Pyrexia (General disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (2)
Feeding disorder (Metabolism and nutrition disorders) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Pneumonia (Infections and infestations) | 5 (9)
Gastroenteritis (Infections and infestations) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Bronchiolitis (Infections and infestations) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2)
Exanthema subitum (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onasemnogene Abeparvovec-xioi (N=33)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Pyrexia (General disorders) | 20 (29)
Crying (General disorders) | 1 (2)
Extravasation (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Necrosis (General disorders) | 1 (1)
Irritability (Psychiatric disorders) | 2 (2)
Nervousness (Psychiatric disorders) | 1 (1)
Psychomotor retardation (Psychiatric disorders) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Stoma site inflammation (Injury, poisoning and procedural complications) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (11)
Aspartate aminotransferase increased (Investigations) | 8 (9)
Oxygen saturation decreased (Investigations) | 2 (2)
Troponin T increased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (2)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Breath sounds (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Haemophilus test positive (Investigations) | 1 (1)
Platelet count increased (Investigations) | 1 (1)
Respiratory syncytial virus test positive (Investigations) | 1 (2)
Respirovirus test positive (Investigations) | 1 (1)
Staphylococcus test positive (Investigations) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (2)
Cyanosis (Cardiac disorders) | 1 (2)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Strabismus (Eye disorders) | 1 (1)
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (15)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 5 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Teething (Gastrointestinal disorders) | 3 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 8 (25)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Device occlusion (Product Issues) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Acne infantile (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (16)
Nasopharyngitis (Infections and infestations) | 4 (8)
Respiratory tract infection (Infections and infestations) | 4 (4)
Ear infection (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3)
Candida infection (Infections and infestations) | 2 (2)
Impetigo (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Bacteriuria (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Dermatitis infected (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Roseola (Infections and infestations) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
A comparison of the results from this study to the results from the natural history observational study (Pediatric Neuromuscular Clinical Research Network (PNCR), Finkel et al, 2014) are included in the Novartis Clinical Trial Results, as a historical control. These full results are available via this link: https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17805.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & has the right to request changes to communications regarding trial results for a period of 30 to 60 days with an additional 6 months, if needed, from the time submitted to the Sponsor for review in order to either remove references to Sponsor's Confidential Information or delay such results communications to permit Sponsor to obtain appropriate Intellectual Property protection as set forth in each of the agreements.

DOCUMENTS (2):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT03461289/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT03461289/SAP_000.pdf